CLINICAL TRIAL: NCT05359991
Title: Revamping Exercise Assessments in Child Health (Project REACH)
Brief Title: Exercise in Child Health
Acronym: Project REACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Children's Hospital of Orange County (Other); Children's Hospital Los Angeles (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Dan Cooper, Professor, University of California, Irvine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20195402
Record Dates: First submitted 2022-03-31; First posted 2022-05-04 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2024-12

CONDITIONS: Cystic Fibrosis; Sickle Cell Disease; SARS CoV 2 Infection
MeSH Terms: conditions — Cystic Fibrosis; Anemia, Sickle Cell; COVID-19 | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Healthy Controls (Active Comparator): Cardiopulmonary Exercise Test (CPET) will be performed to measure cardiorespiratory responses in healthy controls. Exercise will consist of up to 8, 2 minutes bouts of constant work rate cycle ergometry with 1 minute resting intervals between each exercise bout. A subgroup of children will be asked to allow the investigators to obtain blood samples during the exercise session. The following procedures will occur:
  * The child will be in a fasted state.
  * An IV will be placed into the child's arm.
  * Blood sampling will be taken at 4 time points; baseline, and the end of exercise, and at 30 and 60 minutes post exercise.
  Interventions: Other: Exercise
- Children With Documented History of SARS CoV-2 Infection (Experimental): Cardiopulmonary Exercise Test (CPET) will be performed to measure cardiorespiratory responses in children with a documented history of SARS CoV-2 Infection. Exercise will consist of up to 8, 2 minutes bouts of constant work rate cycle ergometry with 1 minute resting intervals between each exercise bout. A subgroup of children will be asked to allow the investigators to obtain blood samples during the exercise session. The following procedures will occur:
  * The child will be in a fasted state.
  * An IV will be placed into the child's arm.
  * Blood sampling will be taken at 4 time points; baseline, and the end of exercise, and at 30 and 60 minutes post exercise.
  Interventions: Other: Exercise
- Children With Sickle Cell Disease (SCD) (Experimental): Cardiopulmonary Exercise Test (CPET) will be performed to measure cardiorespiratory responses in children with Children With Sickle Cell Disease (SCD). Exercise will consist of up to 8, 2 minutes bouts of constant work rate cycle ergometry with 1 minute resting intervals between each exercise bout. A subgroup of children will be asked to allow the investigators to obtain blood samples during the exercise session. The following procedures will occur:
  * The child will be in a fasted state.
  * An IV will be placed into the child's arm.
  * Blood sampling will be taken at 4 time points; baseline, and the end of exercise, and at 30 and 60 minutes post exercise.
  Interventions: Other: Exercise
- Children With Cystic Fibrosis (CF) (Experimental): Cardiopulmonary Exercise Test (CPET) will be performed to measure cardiorespiratory responses in children with Children With Cystic Fibrosis (CF). Exercise will consist of up to 8, 2 minutes bouts of constant work rate cycle ergometry with 1 minute resting intervals between each exercise bout. A subgroup of children will be asked to allow the investigators to obtain blood samples during the exercise session. The following procedures will occur:
  * The child will be in a fasted state.
  * An IV will be placed into the child's arm.
  * Blood sampling will be taken at 4 time points; baseline, and the end of exercise, and at 30 and 60 minutes post exercise.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Cardiopulmonary Exercise Testing (CPET) will be used with Multiple Brief Exercise Bouts (MBEB) in order to obtain the necessary data to yield information on the study outcome variables

SUMMARY:
This study is a cooperative investigation funded by the NIH. The project is a collaboration among three major NIH Clinical Translational Science Awardees: 1) UCI (lead site with its affiliate CHOC), 2) Northwestern University (with its affiliate Lurie Children's Hospital), and 3) USC (with its affiliate Children's Hospital of Los Angeles).

There is an increasing number of children who, through medical advances, now survive diseases and conditions that were once fatal, but which remain chronic and debilitating. A major challenge to improve both the immediate and long term care and health of such children has been the gap in our understanding of how to assess the biological effects of exercise. Like otherwise healthy children, children with chronic diseases and disabilities want to be physically active. The challenge is to determine what constitutes safe and beneficial level of physical activity when the underlying disease or condition [e.g., cystic fibrosis (CF) or sickle cell disease (SCD)] imposes physiological constraints on exercise that are not present in otherwise healthy children. Current exercise testing protocols were based on studies of athletes and high performing healthy individuals and were designed to test limits of performance at very high-intensity, unphysiological, maximal effort. These approaches are not optimal for children and adolescents with disease and disability. This project (REACH-Revamping Exercise Assessment in Child Health) is designed to address this gap. Cohorts of children will be identified with two major genetic diseases (CF and SCD) and measure exercise responses annually as they progress from early puberty to mid or late puberty over a 3-4year period. In addition, in the light of the pandemic, a group of children will be added who were affected by SARS-CoV-2 and investigate their responses to exercise. SARS-CoV-2 has similar long-term symptoms than CF and SCD have. Novel approaches to assessing physiological responses to exercise using advanced data analytics will be examined in relation to metrics of habitual physical activity, circulating biomarkers of inflammation and growth, leukocyte gene expression, and the impact of the underlying CF, SCD or SARS-CoV-2 condition. The data from this study will help to develop a toolkit of innovative metrics for exercise testing that will be made available to the research and clinical community.

DETAILED DESCRIPTION:
New, generalizable approaches are needed for measuring physical fitness and activity across a spectrum of pediatric health and disease.

Exercise in children and adolescents is not merely play but is an essential component of growth and development. Children are among the most spontaneously physically active human beings. It is not surprising that participation in PA (Physical Activity) is a major determinant of health across the lifespan and health-related quality of life in both healthy children and in children with chronic diseases. Despite this essential biologic role for PA, children have not been spared the relentless reduction in levels of PA that is creating a crisis in health care in our nation and throughout the world. Recognition of the enormous morbidity and cost of physical inactivity-related diseases, such as atherosclerosis, type 2 diabetes, and osteoporosis, has spurred new policy initiatives targeting preventive medicine early in life. The concept of pediatric origins of adult health and disease is gaining scientific merit, highlighting the need to transform existing notions of how to evaluate health in a growing child. A physically inactive (even normal weight) child may have no symptoms of disease, but evidence of deterioration in vascular health may already be present. As era of population health management and precision medicine are approaching, the notion of what it means to be a healthy child must change and include robust metrics of physical fitness.

Equally worrisome is that the deleterious health effects of physical inactivity and poor fitness are exacerbated in children with chronic disease and/or disabilities or with environmental-lifestyle conditions like obesity. Children with diseases or conditions previously associated with mortality during the first two decades of life (e.g., SCD, CF) are living longer due to remarkable advances in research and care, but are often unable to achieve levels of PA and fitness associated with health benefits in otherwise healthy children. Not surprisingly, the healthspan [the period of life free from serious chronic diseases and disability of children with chronic diseases is threatened not only by the underlying disease, but by the compounding effects of insufficient PA and sedentary behavior. Increasing PA and fitness is feasible, but has proven quite challenging to implement in a systematic manner. Once a pattern of physical inactivity and a sedentary lifestyle is established, a vicious cycle ensues, in which constraints on PA harm immediate health and contribute to lifelong health impairment ranging from cardiovascular and metabolic disease to osteoporosis. Exactly what constitutes ideal physical fitness in a child with a chronic condition remains unknown. Finding beneficial levels of PA in children with chronic disease or disability is challenging because the optimal range of exercise is much narrower than in a healthy child. Finally, as a result of the COVID-19 pandemic a sizable number of children are experiencing long-term effects such as fatigue, and will be included in our study. Similar to children with CF and SCD, studies of exercise and physical activity will provide insight into disease mechanisms and possible therapies.

ELIGIBILITY:
Inclusion Criteria:

Sickle Cell Disease

* Tanner 1-5, corresponding approximately to ages 10-17 y/o
* SCD diagnosis including all relevant genotypes
* Determined to be in relatively good health as a patient with SCD with no complications from SCD that would render participation the study unadvisable
* No evidence of other disease or disability that would impair participation in PA
* Physician permission to perform CPET
* BMI within the average range for age and condition

Cystic Fibrosis

* Confirmed diagnosis of CF based on either two CF-causing mutations and/or a sweat chloride concentration of > 60 mmol/l after a positive newborn screening test or on two separate occasions
* Tanner 1-5 corresponding approximately to ages 10-17 y/o as documented by a licensed independent provider at screening, or by a validated self-assessment tool
* Determined to be in relatively good health as a patient with CF with no complications from CF that would render participation the study unadvisable as determined by a physician. Examples include history of submassive or massive hemoptysis or moderate to severe pulmonary hypertension.
* BMI in the average range for age and condition
* No evidence of other disease or disability that would impair participation in PA

Comparison (Healthy control)

* Tanner 1-5 corresponding approximately to ages 10-17 y/o
* Determined to be in good health by pre-participation history and physical examination performed by primary care providers or PERC staff
* BMI and PA participation (by history) in the average range for age
* No evidence of disease or disability that would impair participation in PA

Comparison (SARS-CoV-2)

* Tanner 1-5 corresponding approximately to ages 10-17 y/o
* Documented SARS-CoV-2 infection
* Capable of doing exercise as determined by primary care providers or PERC a medical officer

Exclusion Criteria:

Sickle Cell Disease Treatment for substance or alcohol abuse

* Requiring chronic monthly transfusions
* Other conditions that preclude exercise such as neuromotor disease, heart disease, or any other condition that would prevent a child from participating in PA

Cystic Fibrosis Treatment for substance or alcohol abuse

* Other conditions that preclude exercise (such as neuromotor disease, heart disease, or any other condition that would prevent a child from participating in PA)
* FEV1 < 40% predicted based on Global Lung Index equations
* Current infection with Burkholderia cenocepacia or Mycobacterium abscessus

Comparison (Healthy control) Treatment for substance or alcohol abuse or chronic medication use • Determination by PERC staff of unsuitability for exercise

Comparison (SARS-CoV-2) Treatment for substance or alcohol abuse or chronic medication use

• Determination by PERC staff of unsuitability for exercise

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Gas Exchange Variables | 8 Months
  oxygen uptake
Whole Body Lean Mass | 8 Months
  Measured by Dual X-Ray Densitometry
Physical Activity | 8 Months
  Measured by Actigraphy
Biomarkers | 8 Months
  IGF-1
Gene Expression | 8 Months
  Circulating leukocyte gene expression associated with exercise
Gas Exchange Variables | 8 Months
  V̇O2
Gas Exchange Variables | 8 Months
  Carbon dioxide output
Gas Exchange Variables | 8 Months
  V̇CO2
Gas Exchange Variables | 8 Months
  ventilation
Gas Exchange Variables | 8 Months
  V̇E
Gas Exchange Variables | 8 Months
  heart rate (HR)
Fat Mass | 8 Months
  Measured by Dual Energy X-Ray Absorptiometry
% Body Fat | 8 Months
  Measured by Dual X-Ray Densitometry
Whole Body Bone Mineral Content | 8 Months
  Measured by Dual X-Ray Densitometry
Whole Body Bone Mineral Density | 8 Months
  Measured by Dual X-Ray Densitometry
Biomarkers | 8 Months
  IL6
Biomarkers | 8 Months
  C-Reactive Protein
Biomarkers | 8 Months
  Glucose
Biomarkers | 8 Months
  insulin
Biomarkers | 8 Months
  lipid screen
Biomarkers | 8 Months
  lactate
Biomarkers | 8 Months
  CBC
Gene Expression | 8 Months
  Circulating Leukocyte Gene Expression Associated with Sickle Cell Anemia
Gene Expression | 8 Months
  Circulating Leukocyte Gene Expression Associated with Cystic Fibrosis

SECONDARY OUTCOMES:
Behavioral responses to exercise | 8 Months
  PROMIS Parent Fatigue Questionnaire
Standardized assessments | 8 Months
  TANNER Staging Questionnaire
Behavioral responses to exercise | 8 Months
  PROMIS Pediatric Fatigue Questionnaire
Behavioral responses to exercise | 8 Months
  Project REACH NHANES PAQ Adapted Questionnaire
Behavioral responses to exercise | 8 Months
  PEDSQL Fatigue Questionnaire
Behavioral responses to exercise | 8 Months
  Appendices Questionnaire
Standardized assessments | 8 Months
  Block Standardized FFQ

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klentrou P. Influence of Exercise and Training on Critical Stages of Bone Growth and Development. Pediatr Exerc Sci. 2016 May;28(2):178-86. doi: 10.1123/pes.2015-0265. Epub 2016 Feb 17. PMID 26884506
- [Background] Shay CM, Ning H, Daniels SR, Rooks CR, Gidding SS, Lloyd-Jones DM. Status of cardiovascular health in US adolescents: prevalence estimates from the National Health and Nutrition Examination Surveys (NHANES) 2005-2010. Circulation. 2013 Apr 2;127(13):1369-76. doi: 10.1161/CIRCULATIONAHA.113.001559. Epub 2013 Apr 1. PMID 23547177
- [Background] Gates PE, Strain WD, Shore AC. Human endothelial function and microvascular ageing. Exp Physiol. 2009 Mar;94(3):311-6. doi: 10.1113/expphysiol.2008.043349. Epub 2008 Nov 28. PMID 19042980
- [Background] Mielgo-Ayuso J, Aparicio-Ugarriza R, Castillo A, Ruiz E, Avila JM, Aranceta-Batrina J, Gil A, Ortega RM, Serra-Majem L, Varela-Moreiras G, Gonzalez-Gross M. Physical Activity Patterns of the Spanish Population Are Mostly Determined by Sex and Age: Findings in the ANIBES Study. PLoS One. 2016 Feb 25;11(2):e0149969. doi: 10.1371/journal.pone.0149969. eCollection 2016. PMID 26914609
- [Background] Herman KM, Hopman WM, Sabiston CM. Physical activity, screen time and self-rated health and mental health in Canadian adolescents. Prev Med. 2015 Apr;73:112-6. doi: 10.1016/j.ypmed.2015.01.030. Epub 2015 Feb 4. PMID 25660484
- [Background] Maher CA, Toohey M, Ferguson M. Physical activity predicts quality of life and happiness in children and adolescents with cerebral palsy. Disabil Rehabil. 2016;38(9):865-9. doi: 10.3109/09638288.2015.1066450. Epub 2015 Jul 28. PMID 26218617
- [Background] Mutlu EK, Mutlu C, Taskiran H, Ozgen IT. Association of physical activity level with depression, anxiety, and quality of life in children with type 1 diabetes mellitus. J Pediatr Endocrinol Metab. 2015 Nov 1;28(11-12):1273-8. doi: 10.1515/jpem-2015-0082. PMID 26197465
- [Background] Pacheco DR, Silva MJ, Alexandrino AM, Torres RM. Exercise-related quality of life in subjects with asthma: a systematic review. J Asthma. 2012 Jun;49(5):487-95. doi: 10.3109/02770903.2012.680636. Epub 2012 May 3. PMID 22554022
- [Background] Kohl HW 3rd, Craig CL, Lambert EV, Inoue S, Alkandari JR, Leetongin G, Kahlmeier S; Lancet Physical Activity Series Working Group. The pandemic of physical inactivity: global action for public health. Lancet. 2012 Jul 21;380(9838):294-305. doi: 10.1016/S0140-6736(12)60898-8. PMID 22818941
- [Background] Nishi A, Milner DA Jr, Giovannucci EL, Nishihara R, Tan AS, Kawachi I, Ogino S. Integration of molecular pathology, epidemiology and social science for global precision medicine. Expert Rev Mol Diagn. 2016;16(1):11-23. doi: 10.1586/14737159.2016.1115346. Epub 2015 Dec 4. PMID 26636627
- [Background] Briggs AM, Cross MJ, Hoy DG, Sanchez-Riera L, Blyth FM, Woolf AD, March L. Musculoskeletal Health Conditions Represent a Global Threat to Healthy Aging: A Report for the 2015 World Health Organization World Report on Ageing and Health. Gerontologist. 2016 Apr;56 Suppl 2:S243-55. doi: 10.1093/geront/gnw002. PMID 26994264
- [Background] Chu P, Pandya A, Salomon JA, Goldie SJ, Hunink MG. Comparative Effectiveness of Personalized Lifestyle Management Strategies for Cardiovascular Disease Risk Reduction. J Am Heart Assoc. 2016 Mar 29;5(3):e002737. doi: 10.1161/JAHA.115.002737. PMID 27025969
- [Background] Jimenez-Pavon D, Kelly J, Reilly JJ. Associations between objectively measured habitual physical activity and adiposity in children and adolescents: Systematic review. Int J Pediatr Obes. 2010;5(1):3-18. doi: 10.3109/17477160903067601. PMID 19562608
- [Background] Tirakitsoontorn P, Nussbaum E, Moser C, Hill M, Cooper DM. Fitness, acute exercise, and anabolic and catabolic mediators in cystic fibrosis. Am J Respir Crit Care Med. 2001 Oct 15;164(8 Pt 1):1432-7. doi: 10.1164/ajrccm.164.8.2102045. PMID 11704591
- [Background] Alvarado AM, Ward KM, Muntz DS, Thompson AA, Rodeghier M, Fernhall B, Liem RI. Heart rate recovery is impaired after maximal exercise testing in children with sickle cell anemia. J Pediatr. 2015 Feb;166(2):389-93.e1. doi: 10.1016/j.jpeds.2014.10.064. Epub 2014 Dec 2. PMID 25477159
- [Background] Liem RI, Reddy M, Pelligra SA, Savant AP, Fernhall B, Rodeghier M, Thompson AA. Reduced fitness and abnormal cardiopulmonary responses to maximal exercise testing in children and young adults with sickle cell anemia. Physiol Rep. 2015 Apr;3(4):e12338. doi: 10.14814/phy2.12338. PMID 25847915
- [Background] Schneiderman JE, Wilkes DL, Atenafu EG, Nguyen T, Wells GD, Alarie N, Tullis E, Lands LC, Coates AL, Corey M, Ratjen F. Longitudinal relationship between physical activity and lung health in patients with cystic fibrosis. Eur Respir J. 2014 Mar;43(3):817-23. doi: 10.1183/09031936.00055513. Epub 2013 Oct 31. PMID 24176992